CLINICAL TRIAL: NCT02011841
Title: Rifaximin for the Secondary Prevention of Spontaneous Bacterial Peritonitis Recurrence in Cirrhotic Patients: A Prospective, Multicenter, Randomized, Open-label, Controlled Phase III Study
Brief Title: Rifaximin for the Secondary Prevention of Spontaneous Bacterial Peritonitis Recurrence in Cirrhotic Patients
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: We failed to recruit patients
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong-Hoon Lee, Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Rifaximin_SBP
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Spontaneous Bacterial Peritonitis
Keywords: liver cirrhosis; ascites; spontaneous bacterial peritonitis; recurrence
MeSH Terms: conditions — Liver Cirrhosis; Ascites; Recurrence | interventions — Rifaximin; Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rifaximin group (Experimental): Rifaximin 1200 mg/day orally for 6 months
  Interventions: Drug: Rifaximin
- Control group (Active Comparator): Ciprofloxacin 500 mg/day orally for 6 months
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: Rifaximin — rifaximin 1200 mg/day orally for 6 months
  Other Names: Normix
  Arms: Rifaximin group
Drug: Ciprofloxacin — ciprofloxacin 500 mg/day orally for 6 months
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate whether long-term rifaximin administration reduces spontaneous bacterial peritonitis recurrence rate in cirrhotic patients.

DETAILED DESCRIPTION:
* Rifaximin is an antibiotic with a broad-spectrum activity against gram-positive and gram-negative microorganisms, both aerobes and anaerobes within the gastrointestinal tract. The main advantage of rifaximin is that it is poorly absorbable, which minimizes the antimicrobial resistance and adverse events and renders the drug safe in all patient populations. In addition, rifaximin has a better activity against gram-positive organisms than norfloxacin.
* The appreciation of the potential role of enteric flora in the pathogenesis of several gastrointestinal diseases has broadened the clinical use of rifaximin, which is now used for hepatic encephalopathy, small intestine bacterial overgrowth, inflammatory bowel disease, and Clostridium difficile infection. Theoretically, by reducing the total number of the gut bacteria, rifaximin could also be used to achieve intestinal decontamination in patients with liver cirrhosis and ascites, thus preventing spontaneous bacterial peritonitis.
* A small retrospective study concluded that rifaximin suppresses intestinal bacterial overgrowth, bacterial translocation in cirrhotic patients with ascites with no history of previous spontaneous bacterial peritonitis episodes. Prospective clinical trials are warranted to evaluate the role of rifaximin for prevention of spontaneous bacterial peritonitis recurrence in cirrhotic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cirrhosis based on clinical, biochemical, ultrasonographic and/or histological criteria
* Patients who had recovered from an episode of spontaneous bacterial peritonitis
* Age > 18 and <80 years

Exclusion Criteria:

1. Decompensated cirrhotic patients with

   * serum bilirubin > 3.2 mg/dL
   * prothrombin time < 25%
   * serum creatinine > 3 mg/dL
2. Active gastrointestinal bleeding
3. Hepatic encephalopathy > grade 2
4. Patients who have clinical, biochemical or radiological data suggesting hepatocellular carcinoma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The recurrence rate of spontaneous bacterial peritonitis | every 4 weeks, up to 24 weeks
  The proportion of patients who recurred spontaneous bacterial peritonitis.

SECONDARY OUTCOMES:
mortality | up to 24 weeks
  All-cause mortality and cause-specific mortality (mortality due to spontaneous bacterial peritonitis)
The recurrence of culture-negative spontaneous bacterial peritonitis | every 4 weeks, up to 24 weeks
  The proportion of patients who recurred culture-negative spontaneous bacterial peritonitis.
Causative bacteria of recurrent spontaneous bacterial peritonitis | every 4 weeks, up to 24 weeks
  Causative bacteria of recurrent spontaneous bacterial peritonitis and susceptibility
Change of gut microbiota | at baseline, week 12
  Gut microbiota will be analyzed at baseline and week 12
Infections other than spontaneous bacterial peritonitis | every 4 weeks, up to 24 weeks
  Infections other than spontaneous bacterial peritonitis (i.e. urinary tract infection, respiratory tract infection, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Hoon Lee, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea